CLINICAL TRIAL: NCT06830889
Title: A Randomized Controlled Phase Ill Clinical Study of BL-M07D1 for Injection Versus Trastuzumab Emtansine (T-DM1) in the Adjuvant Treatment of HER2-positive Breast Cancer With Residual Invasive Cancer After Neoadjuvant Therapy
Brief Title: A Study of BL-M07D1 Versus T-DM1 in the Adjuvant Treatment of HER2-positive Breast Cancer With Residual Invasive Cancer After Neoadjuvant Therapy
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Collaborators: Baili-Bio (Chengdu) Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BL-M07D1-302
Record Dates: First submitted 2025-02-12; First posted 2025-02-17 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: HER2-positive Breast Cancer
Keywords: HER2-positive breast cancer with residual invasive cancer after neoadjuvant therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BL-M07D1 (Experimental): Participants receive BL-M07D1 as intravenous infusion for the first cycle (3 weeks). Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: BL-M07D1
- T-DM1 (Active Comparator): Participants receive T-DM1 as intravenous infusion for the first cycle (3 weeks). Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: T-DM1

INTERVENTIONS:
Drug: BL-M07D1 — Administration by intravenous infusion for a cycle of 3 weeks.
  Arms: BL-M07D1
Drug: T-DM1 — Administration by intravenous infusion for a cycle of 3 weeks.
  Arms: T-DM1

SUMMARY:
This trial is a registered phase III, randomized, open-label, multicenter study designed to evaluate the efficacy and safety of BL-M07D1 in the adjuvant treatment of HER2-positive breast cancer with residual invasive cancer after neoadjuvant therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent form voluntarily and follow the protocol requirements;
2. Women aged ≥18 years and ≤75 years at the time of written informed consent;
3. Expected survival time ≥6 months;
4. Patients with histologically confirmed HER2-positive invasive breast cancer;
5. Before neoadjuvant therapy, the clinical TNM staging was T1-4, N0-3, M0 (excluding T1N0) based on the 8th edition of the American Joint Committee on Cancer (AJCC) staging system;
6. The presence of residual invasive cancer confirmed by postoperative pathological examination must meet one of the conditions specified in the protocol;
7. Previous neoadjuvant therapy should meet the prescribed treatment conditions;
8. Had received radical mastectomy;
9. Determine hormone receptor (HR) status;
10. The interval between radical surgery and randomization was at least 3 weeks and at most 12 weeks;
11. ECOG score 0 or 1;
12. The toxicity of previous antineoplastic therapy has returned to ≤ grade 1 as defined by NCI-CTCAE v5.0;
13. No blood transfusion within 14 days before the first use of the study drug and no use of colony-stimulating factors were allowed;
14. For premenopausal women with childbearing potential, a pregnancy test must be performed within 7 days before starting treatment, serum pregnancy must be negative, and the patient must not be lactating; All enrolled patients should use adequate and highly effective contraception during the entire treatment cycle and for 7 months after the end of treatment.

Exclusion Criteria:

1. A diagnosis of stage IV metastatic breast cancer was made;
2. Bilateral breast cancer;
3. Any previous history of breast cancer (unilateral or contralateral) except for lobular carcinoma in situ (LCIS);
4. Evidence of clinically significant residual disease or recurrent or metastatic disease after neoadjuvant therapy and surgery;
5. Other primary malignancies diagnosed within 5 years before the first dose;
6. Received previous HER2-ADC, immunotherapy, or other antitumor biological therapy;
7. Subjects are participating in other clinical studies and receiving anti-tumor treatment;
8. Prior treatment with anthracyclines, doxorubicin equivalent cumulative dose > 240 mg/m2; Cumulative dose of epirubicin or liposomal doxorubicin hydrochloride > 480 mg/m2;
9. History of severe cardiovascular or cerebrovascular disease within six months before screening;
10. QT prolongation, complete left bundle branch block, III degree atrioventricular block, frequent and uncontrollable arrhythmia;
11. Poorly controlled hypertension (systolic blood pressure > 150 mmHg or diastolic blood pressure > 100 mmHg);
12. Complicated with pulmonary diseases leading to severe impairment of lung function;
13. A history of ILD/interstitial pneumonia requiring steroid therapy, current ILD/interstitial pneumonia, or suspected such disease during screening; CTCAE v5.0 was used to define grade ≥3 pulmonary disease and grade ≥2 radiation pneumonitis;
14. Human immunodeficiency virus antibody (HIVAb) positive, active hepatitis B virus infection, liver cirrhosis, or hepatitis C virus infection;
15. Had a serious infection within 4 weeks before the first dose of study drug; There was active pulmonary inflammation at the time of screening;
16. Were receiving &gt within 2 weeks before the first dose; 10mg/d prednisone systemic corticosteroids or equivalent anti-inflammatory active drugs or any form of immunosuppressive therapy;
17. Patients with a history of severe allergy to recombinant humanized antibodies or to any of the excipents of BL-M07D1;
18. Known hypersensitivity or delayed hypersensitivity to certain components of T-DM1 or similar drugs, or known contraindications to T-DM1;
19. Had a history of autologous or allogeneic stem cell transplantation or organ transplantation;
20. Have a severe neurological or psychiatric illness;
21. Subjects with clinically significant bleeding or obvious bleeding tendency within 4 weeks before signing the informed consent;
22. Intestinal obstruction, Crohn's disease, ulcerative colitis or chronic diarrhea;
23. Subjects scheduled to receive live vaccine or within 28 days before the first dose;
24. Patients with other serious physical and laboratory abnormalities or poor adherence that may increase the risk of participating in the study, or interfere with the results of the study, and patients who were deemed by the investigators to be unsuitable for participation in the study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 1450 (Estimated)
Dates: Start 2025-06-03 (Actual); Primary Completion 2031-10 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Invasive Disease-free Survival (IDFS) | Up to approximately 77 months
  IDFS refers to the absence of invasive cancer recurrence after breast cancer treatment.

SECONDARY OUTCOMES:
Disease-free Survival(DFS) | Up to approximately 77 months
  DFS is defined as the time from random occurrence of a tumor to recurrence.
Distant Recurrence-free Interval (DRFI) | Up to approximately 77 months
  DRFI is defined as the interval from the date of randomization to the first occurrence of distant recurrence of breast cancer or death due to breast cancer.
Overall Survival (OS) | Up to approximately 77 months
  Overall survival (OS) is defined as the time between the subject's randomization date and subject's death.
Treatment Emergent Adverse Event (TEAE) | Up to approximately 77 months
  TEAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally emerging, or any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition during the treatment of BL-M07D1. The type, frequency and severity of TEAE will be evaluated during the treatment of BL-M07D1.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality